CLINICAL TRIAL: NCT04730986
Title: A Nurse-led, Advance Care Planning Intervention in the Emergency Department: a Pilot Study
Brief Title: A Nurse-led, Advance Care Planning Intervention in the Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Cambia Health Foundation (Other)
Responsible Party: Principal Investigator, Kei Ouchi, Assistant Professor of Emergency Medicine, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2020P002934; K76AG064434 (NIH)
Record Dates: First submitted 2020-12-04; First posted 2021-01-29 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Emergency Department; Motivational Interviewing; Advance Care Planning
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Experimental): This is a single-arm study with all enrolled patients receiving the same ED GOAL Nursing intervention
  Interventions: Behavioral: ED GOAL Nursing

INTERVENTIONS:
Behavioral: ED GOAL Nursing — A brief (<7minutes) interview by an emergency department nurse to empower patients to formulate and communicate their goals for medical care with patients' outpatient clinicians.

SUMMARY:
ED GOAL is a 6-minute, motivational interviewing, advance care planning intervention.

In this study, the investigators will pilot test (Part I) ED GOAL by training research nurses to demonstrate its intervention fidelity and acceptability on older adults with serious illness in the emergency department (ED). Upon demonstrating the intervention fidelity of this intervention in Part I, the investigators will collect patient-centered outcomes (Part II) of 100 older adults with serious illness after leaving the ED. Further in Part III, the investigators will conduct a survey to the participants' outpatient clinicians to find out how to optimize the care coordination from the ED to the outpatient office to facilitate advance care planning conversations.

ELIGIBILITY:
Part 1.

Inclusion Criteria:

* ≥50 years of age AND ≥1 Serious illness* OR ED clinician would not be surprised if patient died in the next 12 months
* English-speaking
* Capacity to consent

Exclusion Criteria:

* Acute physical or emotional distress
* Determined by EM physician not to be appropriate
* Clearly documented goals for medical care** (Unless the treating clinician recommends that the patient needs the intervention)
* Delirium (assessed using 3D-CAM)
* Mild cognitive impairment or dementia (assessed using MiniCog or SBT)
* Already enrolled in this study
* Unable/unwilling to schedule the follow-up outcomes assessment on the calendar.

Part 2.

Inclusion Criteria:

* ≥50 years of age AND ≥1 Serious illness* OR ED clinician would not be surprised if patient died in the next 12 months
* English-speaking
* Patient with mild cognitive impairment or mild dementia with caregiver has a capacity to consent
* Caregivers of patients with moderate/severe dementia has a capacity to consent

Exclusion Criteria:

* Acute physical or emotional distress
* Determined by EM physician not to be appropriate
* Clearly documented goals for medical care** (Unless the treating clinician recommends that the patient needs the intervention)
* Delirium (assessed using 3D-CAM)
* Already enrolled in this study
* Unable/unwilling to schedule the follow-up outcomes assessment on the calendar.

(*NYHA Stage III/IV congestive heart failure, chronic obstructive lung disease on home oxygen, chronic kidney disease on dialysis, or metastatic solid tumor cancer. In addition, patients with NYHA Stage I/II congestive heart failure, chronic obstructive lung disease not on home oxygen, chronic kidney disease not on dialysis, solid tumor cancer without metastasis will be included if recent hospitalization in the last 12 months exists.) (**MOLST, medical order for life-sustaining treatment.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2021-01-29 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Measurement of Intervention Fidelity | Immediately after the the intervention
  Measure the intervention fidelity of ED GOAL Nursing administered by trained research nurses to seriously ill older adults or caregivers of patients with cognitive impairment in the ED (N=30). Trained research nurses will demonstrate intervention fidelity >70% on a prespecified checklist.
Measurement of change in ACP conversations before and after the intervention | Before and one month after the intervention
  Conduct a pre-/post-intervention study (N=100) of ED GOAL Nursing on advance care planning (ACP) conversations one month (28 days) after leaving the ED (confirmed by EMR documentation of new/changes in ACP conversations, advance directive forms, or healthcare proxy, as well as changes in patient's or caregiver's self-reported ACP engagement). ≥25% of participants will have reported completing an ACP conversation, or changed advance directive forms or healthcare proxy, or change in patient's or caregiver's self-reported ACP engagement at one month after leaving the ED.
Identification of key care coordination components from outpatient clinicians. | One month after the intervention
  Conduct a survey on the outpatient clinicians of ED GOAL study participants one month (28 days) after the participating patients leave the ED to identify key care coordination components to maximize the intervention efficacy.

SECONDARY OUTCOMES:
Patient-reported ACP conversation after the intervention | One month after the intervention
  Conduct a survey on the patients to ask if they report having new ACP conversation after the intervention. The outcome is dichotomous (yes or no).
Documentation of new ACP in the electronic health records | Before and one month after the intervention
  Conduct a chart review to find new documentation of advance care planning including new health care proxy form, new medical order for life-sustaining treatment, and new clinicians' free-text documentation of ACP conversations.

CONTACTS AND LOCATIONS:
Overall Officials: Kei Ouchi, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States